CLINICAL TRIAL: NCT04267042
Title: Prospective Double-Cohort Study: Comparing Efficacy of Budesonide Via MAD or INSI in Post-operative Treatment
Brief Title: Comparing Budesonide Via MAD or INSI Prospective Cohort Study
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Amin Javer, Clinical Professor, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H20-00209
Record Dates: First submitted 2020-01-28; First posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps; Allergic Fungal Sinusitis
Keywords: Budesonide; MAD; INSI; CRS; AFRS; Postoperative
MeSH Terms: conditions — Allergic Fungal Sinusitis | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Budesonide via Mucosal Atomization Device (MAD) (Active Comparator): Patients in this arm will administer budesonide using a mucosal atomization device (MAD, Wolfe-Tory Medical, Salt Lake City, UT) once a day at least 5 times a week for 6 months postoperatively. The MAD atomizes the medication into particles from 30-100 um in size thus increasing the surface area for drug absorption.
  Budesonide is provided in nebules (1mg/2cc). Patients will place two nebules of budesonide into the MAD syringe.
  Interventions: Drug: Budesonide; Device: Mucosal Atomization Device
- Budesonide via nasal saline irrigation (INSI) (Active Comparator): Patients in this arm will administer impregnated budesonide in nasal saline irrigation (INSI) using a NeilMed squeeze bottle (NeilMed Pharmaceuticals, Santa Rosa, California) once a day at least 5 times a week for 6 months postoperatively.
  Budesonide is provided in nebules (1mg/2cc).Patients will place two nebules of budesonide into the 240mls of saline.
  Interventions: Drug: Budesonide; Device: NeilMed squeeze bottle for Impregnated Nasal Saline Irrigation

INTERVENTIONS:
Drug: Budesonide — Budesonide is a corticosteroid that is commonly used intranasally to treat CRS.
  Other Names: Pulmicort
Device: Mucosal Atomization Device — MAD is a device used as an addition to a syringe to atomize medication to increase area of distribution. It is used to administer budesonide within the nasal passages and sinuses to administer medication for CRS.
  Other Names: MAD
  Arms: Budesonide via Mucosal Atomization Device (MAD)
Device: NeilMed squeeze bottle for Impregnated Nasal Saline Irrigation — INSI is delivered using a NeilMed squeeze bottle. It is used to administer budesonide within the nasal passages and sinuses to administer medication for CRS.
  Other Names: INSI
  Arms: Budesonide via nasal saline irrigation (INSI)

SUMMARY:
Chronic Rhinosinusitis (CRS) is a common disorder in North America, affecting more than 31 million people annually. Common therapy for CRS includes intranasal corticosteroids (INCS) such as budesonide. At our centre , the current practice is to administer budesonide two ways: the mucosal atomization device (MAD), which is a nasal spray or impregnated budesonide in nasal saline irrigation (INSI), which is a nasal rinse. Our study aims to see which method of administering budesonide has the best treatment outcomes after sinus surgery. This study will follow patients over a six-month period of time.

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) with nasal polyps (CRSwNP) and without nasal polyps (CRSsNP) is a common condition affecting millions of North Americans. CRS is a multifactorial disease that causes inflammation within the sinonasal passages. Symptoms include; dysosmia, nasal blockage, sinus pain, and discolored mucous. Olfactory dysfunction is commonly seen in the CRS patient population. It is estimated that up to 78% of CRS patients have a decreased sense of smell. Therefore, validated smell tests such as Sniffin'Sticks have been used to determine the severity and presence of dysosmia. In addition, patients are frequently colonized with various bacteria or fungi which may further aggravate patient's symptoms. Together, these manifestations lead to a decreased quality of life in CRS patients.

The basis of therapy is to increase mucociliary clearance, improve drainage and relieve obstruction, and eliminate signs of inflammation. Common therapy for the inflamed nasal mucosal lining includes intranasal corticosteroids (INCS) or systemic corticosteroids. Budesonide (Pulmicort) is a corticosteroid which is the mainstay treatment for CRS patients. They have been proven to be very effective in reducing SNOT-22 scores, endoscopic scores, and reducing recurrence in varying severity and subtype of CRS disease.

The current practice at our institution is to administer budesonide via two modalities: the mucosal atomization device (MAD, Wolfe-Tory Medical, Salt Lake City, UT) or impregnated budesonide in nasal saline irrigation (INSI) using a NeilMed squeeze bottle (NeilMed Pharmaceuticals, Santa Rosa, California). The MAD atomizes the medication into particles from 30-100 um in size thus increasing the surface area for drug absorption. At our centre, INSI is frequently employed for CRS patients in the acute postoperative period. Postoperative use of INSI has shown to demonstrate significant improvement in quality of life and endoscopy findings in CRS patients. However, patients can potentially experience headaches and discomfort, which can affect their adherence to this treatment regimen. Therefore, for recalcitrant and non-responsive CRS patients, an alternative treatment method is to utilize budesonide via a MAD in its concentrated form.

Although there is literature that exemplifies the benefit of adding budesonide to postoperative management of CRS patients, there is yet to be a study that assesses the most effective modality of administering the corticosteroid. Therefore, this study aims to prospectively assess the efficacy of INSI and MAD in delivering high-dose nasal corticosteroids in CRS patients. By determining which administration technique is more effective, it will lead to better postoperative outcomes for patients suffering from CRS. Overall, the investigators hope the results from this study will be a step forward in the understanding which administration modality of intranasal corticosteroids is most effective in ameliorating patient disease and quality of life.

Primary Objective:

To compare the postoperative efficacy of budesonide in CRS patients delivered via mucosal atomization device (MAD) or impregnated budesonide in nasal saline irrigation (INSI).

Hypothesis:

The investigators hypothesize that budesonide delivered via MAD will be more effective postoperatively at decreasing objective evidence and subjective symptoms of CRS compared to INSI.

Baseline and Follow-up Visits Evaluation:

The following information will be obtained from each participant

Baseline Demographic data: Age Gender Smoking status

Clinical Data:

* Modified Lund-Kennedy (MLK) scores
* Sinonasal cultures
* Sino-nasal Outcome Test-22 (SNOT-22) and EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) scores
* Sniffin' Sticks Smell Test
* Routine Blood work (Only at week 1 and month 6)

Conduct of Study:

This is a prospective randomized double cohort study at the St. Paul's Sinus Centre. Patients who have an upcoming sinus surgery will be recruited to this study. After the patients have signed the informed consent form and have undergone sinus surgery, they will have their baseline visit. Patients will be divided into the MAD or INSI arm randomly. Patients will be required to take budesonide at least 5 days a week to assure changes seen are directly correlated to taking budesonide. Baseline will be the 1-week postoperative visit following the patient's sinus surgery. Further data will be collected at month 3 and lastly at the patients 6 month follow up visit.

Management of Patient Care

Patients have the right to withdraw from the study at any time. Patients who experience signs and symptoms of hypersensitivity to iodine, burning, itching, pain redness, tiredness, nausea or vomiting will be asked to stop the rinses immediately. The reaction will be noted and the code will be broken so that a discussion can occur between the physician and the patient regarding the use of iodine with the nasal rinses. Patients who meet any of the exclusion criteria that were not noted at the beginning of the study will be removed from this study and the physician will discuss the future management options with the patient.

Sample size:

The investigators expect 60 patients (30 patients per study arm) for the number of participants in this prospective double cohort.

Analysis:

Descriptive statistics will be used to analyze the baseline characteristic data and the data from the administered surveys and objective findings of eosinophil and IgE blood work, cultures, Sniffin' Sticks smell test and MLK scores. In addition, rigorous statistical analysis will be conducted on the Likert scale-based SNOT-22 and EQ-5D-5L surveys. These analyses will include cross-tabulations (Pearson's chi square test) and confidence interval calculations.

Safety Monitoring

Patients who experience signs and symptoms of budesonide reaction will be noted and the code will be broken so that a discussion can occur between the research supervisor and the patient regarding the use of the topical iodine.

Patients can contact the office anytime if they notice any of the signs or symptoms of iodine reaction and will be seen by the research supervisor (or designate) within 24 hours.

Adverse Events (AE's)

All expected and unexpected adverse events will be recorded and graded by the research supervisor. Stable chronic conditions, which are present prior to the clinical trial entry and do not worsen, are not considered adverse events and will be accounted for in the patient's medical history.

Recording/Documentation of Adverse Events

During each patient visit, the research supervisor will ask appropriate questions and perform a physical exam to elicit any adverse events. The research supervisor will also review blood work obtained from the patient. All reportable adverse events will be recorded on appropriate case report form. The research supervisor will also write the stop date, the severity of the AE and his judgment of the AE's relationship to the study.

Serious Adverse Events (SAE's)

An SAE is defined as an AE meeting one of the following:

Death occurring between Day 0 and 182 days (6 months) of the study. Life Threatening Event (defined as a participant at immediate risk of death at the time of the event) In-patient hospitalization or prolongation of existing hospitalization between Day 0 and 42 of the study.

Results in a persistent or significant disability/incapacity In the event of SAE, the research supervisor will discuss with the patient (or next of kin) whether there is a relationship between the study and the SAE. If there is a relationship, the PI will be responsible for coordinating care for the patient until the SAE has been addressed.

Pregnancy During the Trial Patients will be responsible for determining if they are pregnant or become pregnant during the study. If patients notify the PI they are pregnant, they will be removed from the study and the medical management options will be discussed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 19 years and above
* Patients with chronic or recurrent sinusitis (as defined by the American Academy of Otolaryngology) with nasal polyposis or allergic fungal rhinosinusitis
* Patients with an upcoming primary sinus surgery or a revision sinus surgery
* Patients being prescribed INCS for the first time following Functional Endoscopic Sinus Surgery (FESS)

Exclusion Criteria:

* Individuals unable to understand the purpose, methods and conduct of this study
* Patients unwilling to provide informed consent
* Are immuno-compromised, and have impairment in mucociliary function (e.g., cystic fibrosis, Kartagener syndrome)
* Have autoimmune diseases affecting the upper airway (eg Systemic lupus erythematosus, Sjögren's syndrome, systemic sclerosis etc)
* Have sinonasal tumors
* Patients with a history of pituitary disease
* Patients with a known hypersensitivity to cortisol, corticotropin, or cosyntropin
* Recent use of systemic corticosteroids such as prednisone (within last 3 months)
* Patients that are not adherent to budesonide via MAD/INSI treatment
* Patients who are pregnant or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-03 (Estimated); Primary Completion 2021-02-03 (Estimated); Study Completion 2021-02-03 (Estimated)

PRIMARY OUTCOMES:
SNOT-22 questionnaire | 6 months postoperatively
  This is a standard of care form that includes 22 questions about symptoms and social/emotional consequences of your nasal disorder. You will be asked to rate your problems as they have been over the past two weeks. Patients will give a score out of 110 with a higher score relating to worse symptoms.
MLK endoscopic scores | 6 months postoperatively
  This score is based on the endoscopic assessment of polyps, edema, and discharge and are each given score 0-2. A score of 2 indicates a worse outcome.

SECONDARY OUTCOMES:
EQ 5D-5L questionnaireand | 6 months postoperatively
  This is a questionnaire that asks six multiple-choice questions about your mobility, self-care, usual activities, pain/discomfort, anxiety/depression, and overall health.
Sniffin' Sticks Smell tests | 6 months postoperatively
  Many CRS patients have a disturbed/ reduced sense of smell. Sniffn' Sticks is a type of test to assess your sense of smell by using various scented pens. The threshold hold and identification test will be performed. This will give a score out of 32 and a lower score indicates a worse outcome.
Sinus cultures | 6 months postoperatively
  A swab will be taken from your nose to see if there are any bacteria or fungi present.
IgE count | 6 months postoperatively
  Blood will be collected to measure IgE levels.
Eosinophil count | 6 months postoperatively
  Blood will be collected to measure eosinophil levels.

CONTACTS AND LOCATIONS:
Overall Officials: Amin Javer, MD, Principal Investigator — The University of British Columbia and St. Paul's Sinus Centre

IPD SHARING:
Plan to Share IPD: No
We will publish final outcomes as scientific paper.